CLINICAL TRIAL: NCT03575520
Title: A Phase II Study to Evaluate the Safety and Efficacy of Pegteograstim in Korean Breast Cancer Patients Receiving Dose-dense Doxorubicin/Cyclophosphamide
Brief Title: Safety and Efficacy of Pegteograstim in Korean Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0813
Record Dates: First submitted 2018-06-06; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; dose-dense chemotherapy; pegfilgrastim
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim; Doxorubicin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peg group (Experimental)
  Interventions: Drug: Pegfilgrastim; Drug: Doxorubicin/Cyclophosphamide(AC) treatment

INTERVENTIONS:
Drug: Pegfilgrastim — A fixed dose of 6.0 mg pegteograstim was administered subcutaneously on day 2 of each chemotherapy cycle (between 22 and 26 hours after the completion of chemotherapy).
Drug: Doxorubicin/Cyclophosphamide(AC) treatment — doxorubicin 60mg/m2 IV every 2 weeks cyclophosphamide 600mg/m2 IV every 2 weeks
  Four cycles of dose dense AC treatment will be given every 2 weeks.

SUMMARY:
This is a prospective, single arm study, which is examining doxorubicin and cyclophosphamide (AC) once every 2 weeks with pegteograstim support in Korean early breast cancer.

DETAILED DESCRIPTION:
Pegteograstim is a novel monoPEGylated recombinant human G-CSF. In this prospective study, the incidence of febrile neutropenia during four cycles of dose dense (DD) doxorubicin/cyclophosphamide (AC) with pegtoegrastim support is being investigated.

The primary objective of this study is to determine the incidence of febrile neutropenia during four cycles of DD AC with pegteograstim support (8 weeks).

Patients received four cycles of DD-AC (60 mg/m² doxorubicin and 600 mg/m² cyclophosphamide administered intravenously on day 1 every two weeks).

A fixed dose of 6.0 mg pegteograstim was administered subcutaneously on day 2 of each chemotherapy cycle (between 22 and 26 hours after the completion of chemotherapy).

Clinical, hematological, and biochemical assessments were done before the start of each cycle.

Adverse events (AEs) were graded using the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE version 4.03).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of a primary breast cancer (stage I-III)
* Age > 18 years of age and Age < 66 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 1
* Patients who have plan to receive neoadjuvant or adjuvant dose-dense AC chemotherapy
* Adequate organ functions

  1. ANC ≥1500 cells/mm3
  2. PLT ≥100,000 cells/mm3
  3. CCr ≥50 mL/min, or Serum Cr <1.5 x (upper limit of normal, ULN)
  4. Total bilirubin ≤1.5 x ULN
  5. AST (SGOT) ≤2.5 x ULN
  6. ALT (SGPT) ≤2.5 x ULN

Exclusion Criteria:

* Previous chemotherapy history
* Previous bone marrow transplantation history
* Sickle cell anemia
* Radiation therapy within 4 weeks from enrollment
* Previous pegfilgrastim, filgrastim or other colony-stimulating factor treatment within 4 weeks from enrollment
* Clinically significant systemic illness (serious infection, liver, kidney, heart disease)
* Pregnant, breast feeding women

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female population
Enrollment: 63 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
the incidence of febrile neutropenia (FN) | 2months
  FN is defined as neutropenia (<500 neutrophils/μL) with a febrile event (a single oral temperature of ≥38.3°C or a temperature of ≥38.0°C sustained over a one-hour period).

SECONDARY OUTCOMES:
the incidences of febrile neutropenia during the first cycle of chemotherapy | At the end of Cycle 1 (each cycle is 14days)
the incidences of hospitalization for FN | 2months
number of grade 3 or 4 neutropenia in the first cycle of DD-AC | 2months
the incidences of dose delay or reduction of chemotherapy | 2months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Severance Breast Cancer Clinic, Yonsei Cancer Center, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No